CLINICAL TRIAL: NCT05281900
Title: Investigation of Muscular Activation Levels Around the Scapula and Shoulder in Exercises Which Body Weight is Carried on the Arms
Brief Title: Investigation of Muscular Activation Levels Around the Scapula and Shoulder in Exercises Which Body Weight is Carried
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Physical Therapist, PhD, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GO 21/979
Record Dates: First submitted 2021-12-23; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Electromyography; Exercise; Exercise Therapy; Shoulder
Keywords: Electromyography; Exercise; Shoulder
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All participants will complete each stage in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physically active volunteers (Experimental): All volunteers who meet the inclusion criteria will be included in the study.
  Interventions: Diagnostic Test: Clinical Tests; Other: MVIC measurements; Other: Exercises

INTERVENTIONS:
Diagnostic Test: Clinical Tests — Shoulder impingement and instability tests and shoulder normal range of motion measurement.
Other: MVIC measurements — For the normalization of muscle activation during exercises, muscle activation levels during maximum voluntary isometric contraction (MVIC) of the dominant side Upper Trapezius, Middle Trapezius, Lower Trapezius, Serratus Anterior, Biceps Brachii, Triceps Brachii and Infraspinatus muscles will be recorded. Participants will be asked to stop for 10 seconds at the point where they show resistance. A total of three measurements will be taken and the highest value recorded. The areas where the electrodes will be placed will be prepared by shaving and cleaning with alcohol. The electrode placement will be made parallel to the muscle fibers. A rest period of at least 2 minutes will be allowed between measurements.
Other: Exercises — Activation of the scapula and shoulder girdle muscles will be measured during variations of the plank exercise.
  * In the tests, participants will be asked to stay in this position for 10 seconds after providing the standardized stance in the plank position. During the test, a video will be taken and incorrect attempts will be repeated.
  * Determined plank variations will be done in mixed order. Each exercise will be repeated 3 times and the average of the repetitions will be recorded as the result. A 2 minute rest period will be given between exercises.
  * After each exercise, the perceived effort level will be questioned with the BORG scale.
    4 assisted exercises:
    1. Low plank
    2. Low plank w/ isometric shoulder external rotation
    3. High plank
    4. High plank plus
    5. Bear plank
    3 assisted exercises:
    1. Low plank w/ front reach
    2. High plank w/ shoulder taps
    3. High plank w/ toe touch
    2 assisted exercises:
    1. Low plank bird dog
    2. High side plank

SUMMARY:
Closed kinetic chain (CKC) exercises are exercises in which body weight is carried on the distal segment. It is considered advantageous and reliable in many respects compared to open kinetic chain exercises (OKC). For the restoration of functional stability in shoulder rehabilitation, it is recommended to use CKC exercises that carry body weight from the early period. Plank exercise, which is frequently used to strengthen the core area in rehabilitation programs, is performed by transferring weight on the upper extremity. For this reason, it is thought that this exercise will provide an isometric load on the shoulder and scapula muscles. In many previous studies, it has been observed that scapular muscle activations also change with the changes in stability (support surface properties, etc.) in plank exercises and variations in a way that provides a more stable exercise environment. However, as the difficulty level of the used moving floor increased (using softer or unstable surfaces), it was seen that the increase in muscle activation levels was more in favor of the upper trapezius muscle (UT). In a study, it was observed that the UT / Middle Trapeze (MT), UT / Lower Trapezius (LT), UT / Serratus Anterior (SA) ratios were lower in the 3-point supported plank exercise performed on one hand. For this reason, it is thought that while the difficulty level of plank variations is increased in shoulder rehabilitation, body position changes will be more effective in maintaining optimal scapular muscle activation rates instead of using a moving floor. Based on this information, investigating the muscular activation levels for the scapular and shoulder girdle muscles during different variations of the plank exercise in terms of load levels in the targeted muscles will provide valuable information for the management of shoulder exercise programs and post-operative rehabilitation.

It was planned to include 21 healthy physically active individuals between the ages of 18-45 in the study. Muscle activation levels during maximum voluntary isometric contraction (MVIC) of each muscle will be recorded to normalize muscle activation levels during plank variations. Muscle activation levels will be evaluated with a surface electromyography device (Noraxon, Myomotion, USA).

DETAILED DESCRIPTION:
Closed kinetic chain (CKC) exercises are exercises in which body weight is carried on the distal segment. It is considered advantageous and reliable in many respects compared to open kinetic chain exercises (OKC). For the restoration of functional stability in shoulder rehabilitation, it is recommended to use CKC exercises that carry body weight from the early period. Plank exercise, which is frequently used to strengthen the core area in rehabilitation programs, is performed by transferring weight on the upper extremity. For this reason, it is thought that this exercise will provide an isometric load on the shoulder and scapula muscles. In many previous studies, it has been observed that scapular muscle activations also change with the changes in stability (support surface properties, etc.) in plank exercises and variations in a way that provides a more stable exercise environment. However, as the difficulty level of the used moving floor increased (using softer or unstable surfaces), it was seen that the increase in muscle activation levels was more in favor of the upper trapezius muscle (UT). In a study, it was observed that the UT / Middle Trapeze (MT), UT / Lower Trapezius (LT), UT / Serratus Anterior (SA) ratios were lower in the 3-point supported plank exercise performed on one hand. For this reason, it is thought that while the difficulty level of plank variations is increased in shoulder rehabilitation, body position changes will be more effective in maintaining optimal scapular muscle activation rates instead of using a moving floor. Based on this information, investigating the muscular activation levels for the scapular and shoulder girdle muscles during different variations of the plank exercise in terms of load levels in the targeted muscles will provide valuable information for the management of shoulder exercise programs and post-operative rehabilitation.

It was planned to include 21 healthy physically active individuals between the ages of 18-45 in the study. Muscle activation levels during maximum voluntary isometric contraction (MVIC) of each muscle will be recorded to normalize muscle activation levels during plank variations. Muscle activation levels will be evaluated with a surface electromyography device (Noraxon, Myomotion, USA).

ELIGIBILITY:
Inclusion Criteria:

* Physically active participants,
* Having full range of motion of shoulder,
* Having a body mass index less than 30 kg\m2.

Exclusion Criteria:

* Exposure to repetitive overhead shoulder movements due to occupational or sports activities,
* Being symptomatic and positive in at least one of the Hawkins-Kennedy, Neer, Apprehension, Relocation test, Jobe test, and External Rotation Resistance tests,
* Having any injury and/or surgery in the last 6 months,
* Having a current complaint of pain in any part of the body,
* Being diagnosed with a rheumatic, systemic or neurological disease,

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Muscle activation ratio recorded with surface electromyography (sEMG) | 2 hours for each participant
  Electromyography is a measurement method that provides recording and analysis of signals from the central nervous system to the relevant muscle. In this study, muscle activations of the Upper Trapezius(UT), Middle Trapezius(MT), Lower Trapezius(LT), Serratus Anterior(SA), Biceps Brachii(BB), Triceps Brachii(TB) and Infraspinatus(IS) muscles during plank variations will be investigated. Muscle activation levels during maximum voluntary isometric contraction(MVIC) of the muscles will be recorded. The highest value in all repetations of MVIC measurements will be included in the analysis. Muscle activations will be recorded during 10 different plank variations after MVIC measurements. The average value of each repetition will be recorded as a result. As a result of the measurements, %MVIC values of UT, OT, AT, SA, BB, TB, IS, AD muscles and UT/AT, UT/SA, BB/TB, MD/IS activation rates will be calculated in each exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)